CLINICAL TRIAL: NCT05348057
Title: Clinical Study of CMR to Evaluate the Effect of Ivabradine on the Improvement of Left Ventricular Remodeling in STEMI Patients After Primary PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qian geng (Other)
Responsible Party: Sponsor-Investigator, Qian geng, Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: qg-2021-12-01
Record Dates: First submitted 2021-12-05; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine group (Experimental): The starting dose is 5 mg twice a day. After 2 weeks of treatment, if the patient's resting heart rate continues to be higher than 70 beats per minute, increase the dose to 7.5 mg twice a day. If the patient's resting heart rate continues to be less than 50 beats per minute or symptoms related to bradycardia occur, reduce the dose to 2.5 mg
  Interventions: Drug: Ivabradine
- The control group (No Intervention)

INTERVENTIONS:
Drug: Ivabradine — The starting dose is 5 mg twice a day. Adjust the dose according to the actual situation
  Arms: Ivabradine group

SUMMARY:
This study aim to investigate the effect of ivabradine on reducing infarct size and improving left ventricular remodeling after in patients undergoing primary PCI for ST-elevation myocardial infarction through myocardial enhanced MRI.

DETAILED DESCRIPTION:
Investigators will enroll 240 patients with STEMI who were admitted to the Chinese PLA General Hospital between October 2020 and October 2021，the investigators randomly assign eligible patients in a 1:1 ratio to either ivabradine or oral placebo befor primary PCI. The treatment was initiated after primary PCI with ivabradine orally for 6 months. Primary end point of the study was the area of infarct size measured by cardiac magnetic resonance (CMR). Cardiovascular events concluding stroke, repeat revascularization, rehospitalization for acute heart failure, nonfatal myocardial infarction, and all cause death. All adverse clinical events as well as study end points were monitored and adjudicated by the independent event committee.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients: typical chest pain lasting 30 min within the previous 12 h, a clear ST-segment elevation of N0.1 mV in ≥2 contiguous electrocardiographic leads, and elevated blood levels of troponin T
* patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions

Exclusion Criteria:

* had once treated by ivabradine
* history of myocardial infarction
* mechanical complications
* Unable to perform myocardial MRI
* liver and kidney failure
* malignant tumor
* unconscious

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size according to MR delayed enhancement scan | 7 days after PCI
  Two experienced MRI cardiologists analyzed the delayed enhancement image enhancement area of MRI to obtain the area of myocardial infarction through the Segment v1.9 post-processing software
main cardiovascular events | follow up in 6 months
  Acute heart failure, recurrence of myocardial infarction, death from all causes, stroke, cardiac death, recurrent myocardial infarction, recurrent target vascular revascularization, re-admission because of angina pectoris or heart failure

SECONDARY OUTCOMES:
change of the LVEF | follow up in 6 months
  left ventricular ejection fraction (LVEF)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Logeart D, Gueffet JP, Rouzet F, Pousset F, Chavelas C, Solal AC, Jondeau G. Heart rate per se impacts cardiac function in patients with systolic heart failure and pacing: a pilot study. Eur J Heart Fail. 2009 Jan;11(1):53-7. doi: 10.1093/eurjhf/hfn016. PMID 19147457
- [Background] De Ferrari GM, Mazzuero A, Agnesina L, Bertoletti A, Lettino M, Campana C, Schwartz PJ, Tavazzi L. Favourable effects of heart rate reduction with intravenous administration of ivabradine in patients with advanced heart failure. Eur J Heart Fail. 2008 Jun;10(6):550-5. doi: 10.1016/j.ejheart.2008.04.005. Epub 2008 May 16. PMID 18486549
- [Background] Joannides R, Moore N, Iacob M, Compagnon P, Lerebours G, Menard JF, Thuillez C. Comparative effects of ivabradine, a selective heart rate-lowering agent, and propranolol on systemic and cardiac haemodynamics at rest and during exercise. Br J Clin Pharmacol. 2006 Feb;61(2):127-37. doi: 10.1111/j.1365-2125.2005.02544.x. PMID 16433867
- [Background] Ekman I, Chassany O, Komajda M, Bohm M, Borer JS, Ford I, Tavazzi L, Swedberg K. Heart rate reduction with ivabradine and health related quality of life in patients with chronic heart failure: results from the SHIFT study. Eur Heart J. 2011 Oct;32(19):2395-404. doi: 10.1093/eurheartj/ehr343. Epub 2011 Aug 29. PMID 21875859
- [Background] Tardif JC, O'Meara E, Komajda M, Bohm M, Borer JS, Ford I, Tavazzi L, Swedberg K; SHIFT Investigators. Effects of selective heart rate reduction with ivabradine on left ventricular remodelling and function: results from the SHIFT echocardiography substudy. Eur Heart J. 2011 Oct;32(20):2507-15. doi: 10.1093/eurheartj/ehr311. Epub 2011 Aug 29. PMID 21875858
- [Background] Borer JS, Bohm M, Ford I, Komajda M, Tavazzi L, Sendon JL, Alings M, Lopez-de-Sa E, Swedberg K; SHIFT Investigators. Effect of ivabradine on recurrent hospitalization for worsening heart failure in patients with chronic systolic heart failure: the SHIFT Study. Eur Heart J. 2012 Nov;33(22):2813-20. doi: 10.1093/eurheartj/ehs259. Epub 2012 Aug 27. PMID 22927555
- [Background] Borer JS, Bohm M, Ford I, Robertson M, Komajda M, Tavazzi L, Swedberg K; SHIFT Investigators. Efficacy and safety of ivabradine in patients with severe chronic systolic heart failure (from the SHIFT study). Am J Cardiol. 2014 Feb 1;113(3):497-503. doi: 10.1016/j.amjcard.2013.10.033. Epub 2013 Nov 9. PMID 24332674
- [Background] Hidalgo FJ, Anguita M, Castillo JC, Rodriguez S, Pardo L, Duran E, Sanchez JJ, Ferreiro C, Pan M, Mesa D, Delgado M, Ruiz M. Effect of early treatment with ivabradine combined with beta-blockers versus beta-blockers alone in patients hospitalised with heart failure and reduced left ventricular ejection fraction (ETHIC-AHF): A randomised study. Int J Cardiol. 2016 Aug 15;217:7-11. doi: 10.1016/j.ijcard.2016.04.136. Epub 2016 Apr 19. PMID 27167103
- [Background] Sisakian H, Sargsyan T, Khachatryan A. Effect of selective heart rate reduction through sinus node If current inhibition on severely impaired left ventricular diastolic dysfunction in patients with chronic heart failure. Acta Cardiol. 2016 Jun;71(3):317-22. doi: 10.2143/AC.71.3.3152092. No abstract available. PMID 27594127
- [Background] Swedberg K, Komajda M, Bohm M, Borer J, Robertson M, Tavazzi L, Ford I; SHIFT Investigators. Effects on outcomes of heart rate reduction by ivabradine in patients with congestive heart failure: is there an influence of beta-blocker dose?: findings from the SHIFT (Systolic Heart failure treatment with the I(f) inhibitor ivabradine Trial) study. J Am Coll Cardiol. 2012 May 29;59(22):1938-45. doi: 10.1016/j.jacc.2012.01.020. PMID 22617188